CLINICAL TRIAL: NCT05759130
Title: Utility of Sortilin as a Biomarker of Restenosis After Lower Extremity Endovascular Revascularization in a Cohort of Diabetic Patients With Peripheral Artery Disease and Chronic Limb-threatening Ischemia
Brief Title: Utility of Sortilin as a Biomarker of Restenosis After Lower Extremity Endovascular Revascularization
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Flex Andrea, MD, PhD, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 1990
Record Dates: First submitted 2023-02-24; First posted 2023-03-08 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2023-02

CONDITIONS: Peripheral Artery Disease
Keywords: Sortilin; Peripheral Artery Disease; Restenosis; Acute limb ischemia; Amputation; Limb-threatening ischemia
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Sortilin is a 95-kDa protein related to circulating cholesterol. It is found inside different cell types and circulating in blood and it has been associated with the risk of atherosclerosis development and cardiovascular diseases.

The goal of this observational study is to evaluate the potential use of circulating sortilin as a biomarker of vascular adverse outcomes in patients with peripheral artery disease (PAD) and chronic limb-threatening ischemia (CLTI) requiring a procedure of endovascular revascularization.

The main questions it aims to answer are:

* association between sortilin serum levels and risk of restenosis after lower extremity revascularization.
* association between sortilin serum levels and acute limb ischemia, major vascular amputations, and limb-threatening ischemia needing for urgent revascularization after lower extremity revascularization.

Patients with PAD and CLTI requiring lower extremity endovascular revascularization will undergo blood sampling for the dosage of circulating sortilin before the endovascular procedure.

Incidence of restenosis and acute limb ischemia, major vascular amputations, and limb-threatening ischemia needing for urgent revascularization will be collected in a 12-months follow-up and will be associated with sortilin serum levels at baseline.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes mellitus diagnosis;
* Ankle/Brachial Index (ABI) of less than 80;
* at least one lower limb stenosis greater than 50% documented by Ultrasound Color Doppler (US);
* stage 4 or 5 PAD diagnosis according to the Rutherford classification;
* presence of chronic limb threatening ischemia;
* indication for LER of the target arterial stenosis.

Exclusion Criteria:

* statin therapy within the previous 3 months;
* revascularization of the lower limb in the previous 3 months;
* diabetic foot ulcers with signs of active infection or osteomyelitis;
* diabetic peripheral neuropathy;
* homozygous familial hypercholesterolemia;
* absolute contraindication to antiplatelet therapy;
* thrombophilia;
* active cancer;
* active autoimmune disease;
* liver disease at functional status B or C according to Child-Pugh.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We will enroll consecutive statin-naïve subjects with type 2 diabetes mellitus with PAD requiring for endovascular revascularization and admitted to Internal Medicine Cardiovascular Unit of the Fondazione Policlinico Universitario A. Gemelli IRCCS, Roma.
Sampling Method: Probability Sample
Enrollment: 207 (Estimated)
Dates: Start 2019-10-24 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
Correlation between sortilin serum levels before endovascular revascularization and incidence of restenosis | 12-months follow-up
  To evaluate the association between sortilin serum levels before endovascular revascularization and restenosis during the follow-up period.
Correlation between sortilin serum levels before endovascular revascularization and incidence of acute limb ischemia | 12-months follow-up
  To evaluate the association between sortilin serum levels before endovascular revascularization and acute limb ischemia during the follow-up period.
Correlation between sortilin serum levels before endovascular revascularization and incidence of amputations | 12-months follow-up
  To evaluate the association between sortilin serum levels before endovascular revascularization and amputations during the follow-up period.
Correlation between sortilin serum levels before endovascular revascularization and chronic limb-threatening ischemia needing for urgent revascularization | 12-months follow-up
  To evaluate the association between sortilin serum levels before endovascular revascularization and limb-threatening ischemia needing for urgent revascularization during the follow-up period.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Flex, MD, PhD, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, Rome, Italy